CLINICAL TRIAL: NCT05976100
Title: An Open, Simple, Randomized Study of the Safety, Tolerability, Pharmacokinetics of NIOCH-14 in Volunteers Aged 18-50 Years in Parallel Groups
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics of NIOCH-14 in Volunteers Aged 18-50 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Federal Budgetary Research Institution State Research Center of Virology and Biotechnology "Vector" (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIOCH-01/20
Record Dates: First submitted 2023-06-27; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-03

CONDITIONS: Smallpox; Monkeypox; Cowpox; Vaccinia Virus Infection
Keywords: Оrthopoxviruses; Smallpox; NIOCH-14; Сlinical study
MeSH Terms: conditions — Smallpox; Mpox, Monkeypox; Cowpox | interventions — NIOCH-14

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (15 volunteers) (Experimental): Single use:
  Single 200-mg oral dose of NIOCH-14
  Interventions: Drug: NIOCH-14, 200 mg capsule: 1 capsule (200 mg) of NIOCH-14 once orally
- Group 2 (15 volunteers) (Experimental): Single use:
  Single 600-mg oral dose of NIOCH-14
  Interventions: Drug: NIOCH-14, 200 mg capsule: 3 capsules (200 mg each) of NIOCH-14 once orally. (Total 600 mg NIOCH-14 per day)
- Group 3 (15 volunteers) (Experimental): Single use:
  Single 1200-mg oral dose of NIOCH-14 (on the same day in the morning 600 mg and in the evening 600 mg)
  Interventions: Drug: NIOCH-14, 200 mg capsule: 6 capsules (200 mg each) of NIOCH-14 per day orally. (Total 1200 mg NIOCH-14 per day)
- Group 4 (15 volunteers) (Experimental): Multiple application:
  Daily 200-mg oral dose of NIOCH-14 once a day for 6 days
  Interventions: Drug: NIOCH-14, 200 mg capsule: 1 capsule (200 mg) of NIOCH-14 a day orally for 6 days
- Group 5 (15 volunteers) (Experimental): Multiple application:
  Daily 600-mg oral dose of NIOCH-14 once a day for 6 days
  Interventions: Drug: NIOCH-14, 200 mg capsule: 3 capsules (200 mg each) of NIOCH-14 a day orally for 6 days. (Total 600 mg NIOCH-14 per day for 6 days)
- Group 6 (15 volunteers) (Experimental): Multiple application:
  Daily 600-mg oral dose of NIOCH-14 twice a day for 6 days
  Interventions: Drug: NIOCH-14, 200 mg capsule: 3 capsules (200 mg each) of NIOCH-14 twice a day orally for 6 days. (Total 1200 mg NIOCH-14 per day for 6 days)

INTERVENTIONS:
Drug: NIOCH-14, 200 mg capsule: 1 capsule (200 mg) of NIOCH-14 once orally — Volunteers take 1 capsule (200 mg) of NIOCH-14 as a single oral dose.
  Other Names: 7-[N-(4-trifluoromethylbenzoyl)-hydrazinocarbonyl]-tricyclo-[3.2.2.02,4]non-8-en-6-carboxylic acid, 200 mg capsule
  Arms: Group 1 (15 volunteers)
Drug: NIOCH-14, 200 mg capsule: 3 capsules (200 mg each) of NIOCH-14 once orally. (Total 600 mg NIOCH-14 per day) — Volunteers take 3 capsules (200 mg each) of NIOCH-14 as a single oral dose. (Total 600 mg NIOCH-14 per day)
  Other Names: 7-[N-(4-trifluoromethylbenzoyl)-hydrazinocarbonyl]-tricyclo-[3.2.2.02,4]non-8-en-6-carboxylic acid, 200 mg capsule
  Arms: Group 2 (15 volunteers)
Drug: NIOCH-14, 200 mg capsule: 6 capsules (200 mg each) of NIOCH-14 per day orally. (Total 1200 mg NIOCH-14 per day) — Single 1200-mg oral dose. (1200-mg dose of the drug is administered by 600 mg twice a day at 8-00 and 20-00 in the hospital and presence of a clinical investigator or a nurse).
  Other Names: 7-[N-(4-trifluoromethylbenzoyl)-hydrazinocarbonyl]-tricyclo-[3.2.2.02,4]non-8-en-6-carboxylic acid, 200 mg capsule
  Arms: Group 3 (15 volunteers)
Drug: NIOCH-14, 200 mg capsule: 1 capsule (200 mg) of NIOCH-14 a day orally for 6 days — Volunteers take 1 capsule (200 mg) of NIOCH-14 a day orally for 6 days.
  Other Names: 7-[N-(4-trifluoromethylbenzoyl)-hydrazinocarbonyl]-tricyclo-[3.2.2.02,4]non-8-en-6-carboxylic acid, 200 mg capsule
  Arms: Group 4 (15 volunteers)
Drug: NIOCH-14, 200 mg capsule: 3 capsules (200 mg each) of NIOCH-14 a day orally for 6 days. (Total 600 mg NIOCH-14 per day for 6 days) — Volunteers take 3 capsules (200 mg each) of NIOCH-14 a day orally for 6 days.
  Other Names: 7-[N-(4-trifluoromethylbenzoyl)-hydrazinocarbonyl]-tricyclo-[3.2.2.02,4]non-8-en-6-carboxylic acid, 200 mg capsule
  Arms: Group 5 (15 volunteers)
Drug: NIOCH-14, 200 mg capsule: 3 capsules (200 mg each) of NIOCH-14 twice a day orally for 6 days. (Total 1200 mg NIOCH-14 per day for 6 days) — Volunteers take 3 capsules (200 mg each) of NIOCH-14 twice a day orally for 6 days.
  Other Names: 7-[N-(4-trifluoromethylbenzoyl)-hydrazinocarbonyl]-tricyclo-[3.2.2.02,4]non-8-en-6-carboxylic acid, 200 mg capsule
  Arms: Group 6 (15 volunteers)

SUMMARY:
The Aim:

To study safety, tolerability and pharmacokinetics of NIOCH-14 when administered orally using a set of clinical and laboratory-instrumental methods.

The research tasks are to:

* to assess the safety and tolerability of different single doses of the drug;
* to assess the safety and tolerability of different repeated doses of the drug;
* to study pharmacokinetics of single and repeated administration of the drug;
* to assess the data on safety and tolerability to select the optimal drug dosing schedule to resolve the issue of conducting phase II clinical trial in an expanded cohort of volunteers.

DETAILED DESCRIPTION:
An open, simple, randomized study of the safety, tolerability, and pharmacokinetics of NIOCH-14 in volunteers aged 18-50 years in parallel groups will be conducted.

The study included 90 healthy volunteers of both sexes aged 18-50 years who met the inclusion criteria, had no exclusion criteria and underwent all screening procedures.

Grouping of the volunteers:

1) For a single dose of the drug, three groups will be formed: group 1 - 15 volunteers, single 200-mg oral dose; group 2 - 15 volunteers, single 600-mg oral dose; group 3 - 15 volunteers, single 1200-mg oral dose. Before drug administration, volunteers should be hospitalized for a day in the hospital of Federal State Budgetary Healthcare Institution "Medical and Sanitary Unit No. 163 of the Federal Medical and Biological Agency" (FGBUZ MSCH-163, FMBA Russia).

The drug will be first given to 5 healthy volunteers in Group 1. The volunteers will be followed up daily by a clinical investigator for 7 days. In the absence of changes in clinical analyzes and adverse events and the approval of the findings by the IDMC, the remaining subjects in Group 1 will begin to receive the drug.

After 7 days of the follow-up, the first 5 volunteers in Group 2 (600 mg) will start receiving the drug. After 7 days, the remaining 10 volunteers in Group 2 will receive the drug.

The first 5 volunteers in Group 3 will start receiving the drug after obtaining the results for the volunteers in Group 2.

If the volunteers feel satisfactory, they will be discharged on the 2nd day, and then will have to visit the clinical site for examination and identification of adverse events daily for 7 days, after which all volunteers will be given self- monitoring diaries for self-completion to record all adverse events. The volunteers have to present for examination and clinical testing on the 10th, 20th, 30th and 90th day after receiving the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent of a volunteer to participate in the clinical study, obtained prior to any of the study procedures.
2. A verified diagnosis "healthy" based on findings of standard clinical, laboratory and instrumental methods of examination.
3. Age from 18 to 50 years inclusive.
4. Body mass index from 18.5 to 30 kg/m3.
5. Ability to attend all scheduled visits and all scheduled procedures and examinations.
6. Consent of volunteers to use effective methods of contraception throughout the study.

Exclusion Criteria:

1. Known hypersensitivity to any component of the studied drug.
2. Aggravated history of allergies.
3. Drug intolerance.
4. Pregnancy and the period of breastfeeding.
5. Military personnel.
6. Persons in custody in pre-trial detention centers and serving sentences in penitentiaries.
7. Children's age under 18.
8. Acute infectious diseases less than 4 weeks before the start of the study.
9. Acute or chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine system, as well as diseases of the gastrointestinal tract, liver, blood, kidneys, surgical interventions to the gastrointestinal tract (with the exception of appendectomy).
10. Immunosuppressive conditions: congenital or acquired immunodeficiency syndrome (including HIV infection), leukemia, malignant tumors, organ transplantation, cellular and humoral immunodeficiencies.
11. Immunosuppressive therapy: treatment with antimetabolites, high doses of corticosteroids for 14 days or more, radio and x-ray therapy, etc.
12. Regular medication intake less than 2 weeks prior to the start of the study.
13. Taking medications that have a pronounced effect on hemodynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, etc.) less than 30 days before the start of the study.
14. Donation (450 ml of blood or plasma or more) less than 2 months before the start of the study.
15. Participation in other clinical trials less than 3 months prior to study enrollment.
16. Drinking more than 10 units of alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml of wine or 50 ml of alcohol) or a history of alcoholism, drug addiction, drug abuse.
17. Smoking of more than 10 cigarettes a day.
18. Failure to meet inclusion criteria.
19. Premenopausal women (last menstrual period ≤ 1 year prior to signing of informed consent) who are not surgically sterile.
20. Women with a childbearing potential not using or planning to use acceptable means of contraception during the study and give no consent to urine pregnancy testing during the study. Acceptable means of contraception include ectopic devices, oral, implanted, or injectable contraceptives.
21. Nervous and mental diseases: central nervous system (CNS) traumas with residual effects, encephalitis and encephalomyelitis (including post-vaccination), meningitis, polyradiculoneuritis (including a history of polyradiculoneuritis), epilepsy, hydrocephalus in the stage of decompensation or subcompensation, demyelinating and degenerative nervous system damage (muscle degeneration, etc.), stroke; compensated hydrocephalus, Down's disease, Little's disease, CNS damage without residual effects, history of febrile convulsions, mental illnesses.

Early (premature) exclusion of subjects from the study (reasons for discontinuation of the studied drug administration):

After randomization and the start of the clinical phase, a clinical investigator may exclude a subject early from the study if:

* The decision of the clinical investigator to exclude a volunteer is in the best interests of the volunteer.
* Erroneous inclusion (inclusion and non-inclusion criteria were not allowed for) or the appearance of non-inclusion criteria during the study.
* Investigator's or Client's decision to exclude a volunteer from the study due to a clinically significant protocol deviation/violation of the protocol.
* Any adverse event requiring the prescription of drugs that are not permitted by the protocol of the study (exacerbation of chronic diseases of the liver, kidneys, pancreas, heart; occurrence of infectious (influenza and other acute respiratory viral infections, tonsillitis, hepatitis, etc.) or oncological diseases during the study.
* Volunteer's refusal to continue participation in the study or his indiscipline.
* Volunteer's desire to terminate the study early for any reason.
* Failure of a volunteer to attend a scheduled visit without notifying the clinical investigator, and loss of communication with a volunteer.
* Positive urine drug test and/or alcohol breath test at visits.
* Pregnancy. Identification of reasons for premature termination of the study in enrolled subjects leads to their exclusion from the study at the stage when these reasons were identified. In each case of premature termination of the study by a volunteer/exclusion of a volunteer from the study, the clinical investigator must make an appropriate entry in the Individual Registration Card (IRC) with the obligatory indication of the reason for the premature termination or exclusion of a volunteer from the study, and inform the authorized representative of the Customer.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Monitoring of erythrocyte level (in clinical (general) blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a clinical (general) blood test is performed: erythrocyte level is measured (10^12 pcs/l). Value changes between time points are calculated.
Monitoring of leukocyte level (in clinical (general) blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a clinical (general) blood test is performed: leukocyte level is measured (10⁹ pcs/l). Value changes between time points are calculated.
Monitoring of platelet level (in clinical (general) blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a clinical (general) blood test is performed: platelet level is measured (10⁹ pcs/l). Value changes between time points are calculated.
Monitoring of hemoglobin level (in clinical (general) blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a clinical (general) blood test is performed: hemoglobin level is measured (g/l). Value changes between time points are calculated.
Monitoring of erythrocyte sedimentation rate (ESR) (in clinical (general) blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a clinical (general) blood test is performed: ESR is measured (mm/hr). Value changes between time points are calculated.
Monitoring of stab neutrophil level (in clinical (general) blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a clinical (general) blood test is performed: stab neutrophil level is measured (%). Value changes between time points are calculated.
Monitoring of segmented neutrophil level (in clinical (general) blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a clinical (general) blood test is performed: segmented neutrophil level is measured (%). Value changes between time points are calculated.
Monitoring of eosinophil level (in clinical (general) blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a clinical (general) blood test is performed: eosinophil level is measured (%). Value changes between time points are calculated.
Monitoring of basophil level (in clinical (general) blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a clinical (general) blood test is performed: basophil level is measured (%). Value changes between time points are calculated.
  10. Monitoring of monocyte level (in clinical (general) blood test).
Monitoring of monocyte level (in clinical (general) blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a clinical (general) blood test is performed: monocyte level is measured (%). Value changes between time points are calculated.
Monitoring of lymphocyte level (in clinical (general) blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a clinical (general) blood test is performed: lymphocyte level is measured (%). Value changes between time points are calculated.
Monitoring of alanine transaminase activity (in biochemical blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a biochemical blood test is performed: the activity of alanine transaminase is measured (U/l). Value changes between time points are calculated.
Monitoring of aspartate aminotransferase activity (in biochemical blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a biochemical blood test is performed: the activity of aspartate aminotransferase is measured (U/l). Value changes between time points are calculated.
Monitoring of alkaline phosphatase activity (in biochemical blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a biochemical blood test is performed: the activity of alkaline phosphatase is measured (U/l). Value changes between time points are calculated.
Monitoring of total protein level (in biochemical blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a biochemical blood test is performed: total protein level is measured (g/l). Value changes between time points are calculated.
Monitoring of total bilirubin level (in biochemical blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a biochemical blood test is performed: total bilirubin level is measured (μmol/l). Value changes between time points are calculated.
Monitoring of glucose level (in biochemical blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a biochemical blood test is performed: glucose level is measured (μmol/l). Value changes between time points are calculated.
Monitoring of creatinine level (in biochemical blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a biochemical blood test is performed: creatinine level is measured (μmol/l). Value changes between time points are calculated.
Monitoring of urea level (in biochemical blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a biochemical blood test is performed: urea level is measured (μmol/l). Value changes between time points are calculated.
Monitoring of thymol test values (in biochemical blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a biochemical blood test is performed: thymol test value is measured (S-H). Value changes between time points are calculated
Monitoring of C-reactive protein (CRP) level (in biochemical blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a biochemical blood test is performed: CRP level is measured (mg/ml). Value changes between time points are calculated.
Monitoring of prothrombin index (PTI) (in biochemical blood test). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a biochemical blood test is performed: PTI is measured (%). Value changes between time points are calculated.
Monitoring of urine color (in common urine analysis). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a common urine analysis is performed: urine color is assessed. Urine color changes between time points are evaluated.
Monitoring of urine transparency (in common urine analysis). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a common urine analysis is performed: urine transparency is assessed.
  Urine transparency changes between time points are evaluated.
Monitoring of urine pH (in common urine analysis). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a common urine analysis is performed: urine pH is measured. Urine pH changes between time points are calculated.
Monitoring of urine specific density (in common urine analysis). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a common urine analysis is performed: urine specific density is measured.
  Urine specific density changes between time points are calculated.
Monitoring of protein level (in common urine analysis). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a common urine analysis is performed: protein level (g/l) is measured.
  Value changes between time points are calculated.
Monitoring of glucose level (in common urine analysis). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a common urine analysis is performed: glucose level (μmol/l) is measured.
  Value changes between time points are calculated.
Monitoring of leukocyte level (in common urine analysis). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a common urine analysis is performed: leukocyte level (10⁹/l) is measured.
  Value changes between time points are calculated.
Monitoring of erythrocyte level (in common urine analysis). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a common urine analysis is performed: erythrocyte level (10^12 /l) is measured. Value changes between time points are calculated.
Monitoring of bacteria (in common urine analysis). | Groups 1-6: at days 0, 3, 7, 10, 20, 30, 90.
  On control days, a common urine analysis is performed: bacterial number (units per field) is measured.
  Value changes between time points are calculated.
Monitoring for the occurrence of adverse events and serious adverse events at least likely related to the studied drug during the study. | Groups 1-6: at days 2-10, 20, 30, 90.
  At each visit, the occurrence of adverse events and serious adverse events, at least likely related to the studied drug, is monitored. The change in the volunteer's state between time points is evaluated.
Monitoring for the occurrence of any adverse events during the study. | Groups 1-6: at days 2-10, 20, 30, 90.
  At each visit, the incidence of any adverse events is measured. The change in the volunteer's state between time points is evaluated.
Monitoring for the occurrence of any serious adverse events during the study. | Groups 1-6: at days 2-10, 20, 30, 90.
  At each visit, the incidence of any serious adverse events that lead to the exclusion of participant from the study is measured. The change in the volunteer's state between time points is evaluated.
Monitoring of body temperature at regular intervals. | Groups 1-6: at days 0, 1-10, 20, 30, 90.
  Body temperature is recorded (degrees Celsius, °C) on control days. Changes in the values of this parameter between time points are calculated.
Monitoring of blood pressure at regular intervals. | Groups 1-6: at days 0, 1-10, 20, 30, 90.
  Systolic and diastolic blood pressure is recorded (mm Hg). Changes in the values of this parameter between time points are calculated.
Monitoring of heart rate at specified intervals. | Groups 1-6: at days 0, 1-10, 20, 30, 90.
  Heart rate is recorded (beats per minute) on control days. Changes in the values of this parameter between time points are calculated.
Monitoring of respiratory movement frequency at specified intervals. | Groups 1-6: at days 0, 1-10, 20, 30, 90.
  On the control days, the frequency of respiratory movements (per minute) is recorded. Changes in the values of this parameter between time points are calculated.
Electrocardiography findings (ECG). | Groups 1-6: at days 0, 1, 3, 7.
  On control days, a planned standard 12-lead ECG is performed (with measurement of heart rate [HR], PR, QRS, QT intervals and QTc calculation). It is performed in the supine position after 5 minutes of rest. The rhythm record in the respective leads must contain measurable data for at least three cardiac cycles. Changes in the values between time points are calculated.
  If there are any changes in the ECG, the clinical investigator should evaluate their clinical significance.

SECONDARY OUTCOMES:
Abdominal ultrasound findings. | Groups 1-6: at days 0, 7.
  On control days, the absence of signs of abdominal organ changes is monitored using ultrasound.
  Changes in the values between time points are calculated.
Monitoring of the pharmacokinetic parameter "Cmax" for ST-246 (active metabolite of NIOCH-14) | Groups 1-3: at days 1-5; groups 4-6: at days 1-10.
  On control days, blood concentration of the active NIOCH-14 metabolite, namely ST-246, is determined using mass spectrometry. The maximum concentration of a substance in the blood plasma, achieved after substance absorption (pharmacokinetic parameter Cmax) is measured. Changes in the values of this parameter between time points are calculated.
Monitoring of the pharmacokinetic parameter "Tmax" for ST-246 (active metabolite of NIOCH-14) | Groups 1-3: at days 1-5; groups 4-6: at days 1-10.
  On control days, blood concentration of the active NIOCH-14 metabolite, namely ST-246, is determined using mass spectrometry. The pharmacokinetic parameter Tmax (the time point when the maximum concentration of a substance in the blood is reached) is measured. Changes in the values of this parameter between time points are calculated.
Monitoring of the pharmacokinetic parameter "Cmax /AUC" for ST-246 (active metabolite of NIOCH-14) | Groups 1-3: at days 1-5; groups 4-6: at days 1-10.
  On control days, blood concentration of the active NIOCH-14 metabolite, namely ST-246, is determined using mass spectrometry. The pharmacokinetic parameter "Cmax /AUC" (the rate of substance entry into the systemic circulation from the injection site) is measured. Changes in the values of this parameter between time points are calculated.
Monitoring of the pharmacokinetic parameter "Elimination rate" for ST-246 (active metabolite of NIOCH-14) | Groups 1-3: at days 1-5; groups 4-6: at days 1-10.
  On control days, blood concentration of the active NIOCH-14 metabolite, namely ST-246, is determined using mass spectrometry. The pharmacokinetic parameter "Elimination rate" (the rate of substance elimination from systemic circulation through biotransformation (metabolism) in the body, and excretion) is measured. Changes in the values of this parameter between time points are calculated.
Monitoring of the pharmacokinetic parameter "T½" for ST-246 (active metabolite of NIOCH-14) | Groups 1-3: at days 1-5; groups 4-6: at days 1-10.
  On control days, blood concentration of the active NIOCH-14 metabolite, namely ST-246, is determined using mass spectrometry. The pharmacokinetic parameter "T½" (half-life, the time of 50% substance concentration reduction in plasma) is measured. Changes in the values of this parameter between time points are calculated.
Monitoring of the pharmacokinetic parameter "AUC" for ST-246 (active metabolite of NIOCH-14) | Groups 1-3: at days 1-5; groups 4-6: at days 1-10.
  On control days, blood concentration of the active NIOCH-14 metabolite, namely ST-246, is determined using mass spectrometry. The pharmacokinetic parameter "AUC" (area under the curve. It is the integral parameter that characterizes the total amount of a substance entering the blood) is measured. Changes in the values of this parameter between time points are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I. Kuzubov, PhD, Principal Investigator — FGBUZ MSCH-163, FMBA Russia
Locations (1):
- Federal State Budgetary Healthcare Institution - Medical and Sanitary Unit No. 163 of the Federal Medical and Biological Agency (FGBUZ MSCH-163, FMBA Russia), Novosibirsk, Koltsovo, Novosibirsk Region, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campe H, Zimmermann P, Glos K, Bayer M, Bergemann H, Dreweck C, Graf P, Weber BK, Meyer H, Buttner M, Busch U, Sing A. Cowpox virus transmission from pet rats to humans, Germany. Emerg Infect Dis. 2009 May;15(5):777-80. doi: 10.3201/eid1505.090159. PMID 19402967
- [Background] Ladnyi I.D. Eradication of Smallpox and Prevention of Its Recurrence. - Moscow: Meditsina, 1985. - 224 P.
- [Background] Fenner F., Henderson D.A., Arita I., et al. Smallpox and its eradication. - Geneva: World Health Organization, 1988.
- [Background] Scientific review of variola virus research, 1999-2010//WHO/HSE/GAR/BDP/2010.3. December 2010
- [Background] Borisevich SV, Marennikova SS, Makhlay AA, Terent'ev AI, Loginova SY, Perekrest VV, Krasnyanskiy VP, Bondarev VP, Rybak SI Cowpox: spread features after the abolition of mandatory smallpox vaccination. Journal of microbiology, epidemiology and immunobiology. 2012; N. 3. 103-107.
- [Background] Hemmer CJ, Littmann M, Lobermann M, Meyer H, Petschaelis A, Reisinger EC. Human cowpox virus infection acquired from a circus elephant in Germany. Int J Infect Dis. 2010 Sep;14 Suppl 3:e338-40. doi: 10.1016/j.ijid.2010.03.005. Epub 2010 Jun 26. PMID 20580588
- [Background] Ninove L, Domart Y, Vervel C, Voinot C, Salez N, Raoult D, Meyer H, Capek I, Zandotti C, Charrel RN. Cowpox virus transmission from pet rats to humans, France. Emerg Infect Dis. 2009 May;15(5):781-4. doi: 10.3201/eid1505.090235. PMID 19402968
- [Background] Baran V.M., Zubritsky P.K. Human cowpox. Healthcare (Minsk). 1997; No. 3. P. 40
- [Background] Marennikova SS, Gashnikov PV, Zhukova OA, Riabchikova EI, Strel'tsov VV, Riazankina OI, Chekunova EV, Ianova NN, Shchelkunov SN. [The biotype and genetic characteristics of an isolate of the cowpox virus causing infection in a child]. Zh Mikrobiol Epidemiol Immunobiol. 1996 Jul-Aug;(4):6-10. Russian. PMID 9027179
- [Background] Shchelkunov SN. Emergence and reemergence of smallpox: the need for development of a new generation smallpox vaccine. Vaccine. 2011 Dec 30;29 Suppl 4:D49-53. doi: 10.1016/j.vaccine.2011.05.037. Epub 2011 Dec 18. PMID 22185833
- [Background] Shchelkunov SN. An increasing danger of zoonotic orthopoxvirus infections. PLoS Pathog. 2013;9(12):e1003756. doi: 10.1371/journal.ppat.1003756. Epub 2013 Dec 5. PMID 24339772
- [Background] Marennikova S.S., Shchelkunov S.N. Orthopoxviruses pathogenic to humans. M.: KMK Scientific Press Ltd. - 1998. - 385 P.
- [Background] Onishchenko GG, Sandkhchiev LS, Netesov SV, Shchelkunov SV. [Bioterrorism: national and global threats]. Zh Mikrobiol Epidemiol Immunobiol. 2000 Nov-Dec;(6):83-5. No abstract available. Russian. PMID 11210651
- [Background] Yang G, Pevear DC, Davies MH, Collett MS, Bailey T, Rippen S, Barone L, Burns C, Rhodes G, Tohan S, Huggins JW, Baker RO, Buller RL, Touchette E, Waller K, Schriewer J, Neyts J, DeClercq E, Jones K, Hruby D, Jordan R. An orally bioavailable antipoxvirus compound (ST-246) inhibits extracellular virus formation and protects mice from lethal orthopoxvirus Challenge. J Virol. 2005 Oct;79(20):13139-49. doi: 10.1128/JVI.79.20.13139-13149.2005. PMID 16189015
- [Background] Burgasov P.N., Nikolaevsky G.P. Smallpox. - M.: Medicine, 1972. - 207 P.
- [Background] Mazurkov OY, Kabanov AS, Shishkina LN, Sergeev AA, Skarnovich MO, Bormotov NI, Skarnovich MA, Ovchinnikova AS, Titova KA, Galahova DO, Bulychev LE, Sergeev AA, Taranov OS, Selivanov BA, Tikhonov AY, Zavjalov EL, Agafonov AP, Sergeev AN. New effective chemically synthesized anti-smallpox compound NIOCH-14. J Gen Virol. 2016 May;97(5):1229-1239. doi: 10.1099/jgv.0.000422. Epub 2016 Feb 8. PMID 26861777
- [Background] Mazurkov OY, Shishkina LN, Bormotov NI, Skarnovich MO, Serova OA, Mazurkova NA, Chernonosov AA, Tikhonov AY, Selivanov BA. Estimation of Absolute Bioavailability of the Chemical Substance of the Anti-Smallpox Preparation NIOCH-14 in Mice. Bull Exp Biol Med. 2020 Dec;170(2):207-210. doi: 10.1007/s10517-020-05034-x. Epub 2020 Dec 2. PMID 33263846
- [Background] Selivanov B.A., et al. 7-[N'-(4-trifluoromethylbenzoyl)-hydrazinocarbonyl]-tricyclo[3.2.2.02,4]non-8-ene-6-carboxylic acid, having antiviral activity. Patent RU No. 2412160, publ. 20.02.2011, Bull. No. 5.
- [Background] Shishkina L.N., Sergeev A.N., Agafonov A.P., Sergeev A.A., Kabanov A.S., Bulychev L.E., Sergeev A.A., Galakhova D.O., Pyankov O.V., Bormotov N.I., Shchukin G.I., Selivanov B.A., Tikhonov A.Ya. Medicated product for smallpox virus and method for producing and using it. Patent RU No. 2543338, publ. 02/27/2015, Bulletin No. 6.
- [Background] Chen Y, Amantana A, Tyavanagimatt SR, Zima D, Yan XS, Kasi G, Weeks M, Stone MA, Weimers WC, Samuel P, Tan Y, Jones KF, Lee DR, Kickner SS, Saville BM, Lauzon M, McIntyre A, Honeychurch KM, Jordan R, Hruby DE, Leeds JM. Comparison of the safety and pharmacokinetics of ST-246(R) after i.v. infusion or oral administration in mice, rabbits and monkeys. PLoS One. 2011;6(8):e23237. doi: 10.1371/journal.pone.0023237. Epub 2011 Aug 15. PMID 21858040
- [Background] van Gerven J, Bonelli M. Commentary on the EMA Guideline on strategies to identify and mitigate risks for first-in-human and early clinical trials with investigational medicinal products. Br J Clin Pharmacol. 2018 Jul;84(7):1401-1409. doi: 10.1111/bcp.13550. Epub 2018 May 30. No abstract available. PMID 29451320